CLINICAL TRIAL: NCT02960906
Title: A Phase 2 BIOmarker Driven Trial With Nivolumab and Ipilimumab or VEGFR tKi in Naïve Metastatic Kidney Cancer
Brief Title: A BIOmarker Driven Trial With Nivolumab and Ipilimumab or VEGFR tKi in Naïve Metastatic Kidney Cancer
Acronym: BIONIKK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Association Pour La Recherche des Thérapeutiques Innovantes en Cancérologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIONIKK
Record Dates: First submitted 2016-08-18; First posted 2016-11-10 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Clear Cell Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — Nivolumab; Ipilimumab; pazopanib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- ccRCC molecular subgroup 1: 1A (Experimental): ccRCC molecular subgroup 1 -> randomisation: subjects with ccRCC1 treated with nivolumab 240mg IV every 2 weeks until disease progression, unacceptable toxicity or other reasons specified in the protocol.
  Starting from the Cycle 7 possibility to switch from nivolumab 240 mg every 2 weeks to 480 mg every 4 weeks according to the Investigator's preference.
  Interventions: Drug: Nivolumab
- ccRCC molecular subgroup 1: 1B (Experimental): ccRCC molecular subgroup 1 -> randomisation: subjects with ccRCC1 treated with nivolumab 3 mg/kg IV combined with ipilimumab 1 mg/kg IV every 3 weeks for 4 doses then nivolumab 240mg IV every 2 weeks until disease progression, unacceptable toxicity or other reasons specified in the protocol.
  Starting from the Cycle 7 possibility to switch from nivolumab 240 mg every 2 weeks to 480 mg every 4 weeks according to the Investigator's preference.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- ccRCC molecular subgroup 4: 4A (Experimental): ccRCC molecular subgroup 4 -> randomisation: subjects with ccRCC1 treated with nivolumab 240mg IV every 2 weeks until disease progression, unacceptable toxicity or other reasons specified in the protocol.
  Starting from the Cycle 7 possibility to switch from nivolumab 240 mg every 2 weeks to 480 mg every 4 weeks according to the Investigator's preference.
  Interventions: Drug: Nivolumab
- ccRCC molecular subgroup 4: 4B (Experimental): ccRCC molecular subgroup 4 -> randomisation: subjects with ccRCC1 treated with nivolumab 3 mg/kg IV combined with ipilimumab 1 mg/kg IV every 3 weeks for 4 doses then nivolumab 240mg IV every 2 weeks until disease progression, unacceptable toxicity or other reasons specified in the protocol.
  Starting from the Cycle 7 possibility to switch from nivolumab 240 mg every 2 weeks to 480 mg every 4 weeks according to the Investigator's preference.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- ccRCC molecular subgroup 2: 2C (Experimental): ccRCC molecular subgroup 2 -> randomisation: TKI (sunitinib 50mg daily or Pazopanib 800mg daily) according to investigator's choice until disease progression, unacceptable toxicity or other reasons specified in the protocol.
  Interventions: Drug: Pazopanib; Drug: Sunitinib
- ccRCC molecular subgroup 2: 2B (Experimental): ccRCC molecular subgroup 2 -> randomisation: subjects with ccRCC1 treated with nivolumab 3 mg/kg IV combined with ipilimumab 1 mg/kg IV every 3 weeks for 4 doses then nivolumab 240mg IV every 2 weeks until disease progression, unacceptable toxicity or other reasons specified in the protocol.
  Starting from the Cycle 7 possibility to switch from nivolumab 240 mg every 2 weeks to 480 mg every 4 weeks according to the Investigator's preference.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- ccRCC molecular subgroup 3: 3B (Experimental): ccRCC molecular subgroup 3 -> randomisation: subjects with ccRCC1 treated with nivolumab 3 mg/kg IV combined with ipilimumab 1 mg/kg IV every 3 weeks for 4 doses then nivolumab 240mg IV every 2 weeks until disease progression, unacceptable toxicity or other reasons specified in the protocol.
  Starting from the Cycle 7 possibility to switch from nivolumab 240 mg every 2 weeks to 480 mg every 4 weeks according to the Investigator's preference.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- ccRCC molecular subgroup 3: 3C (Experimental): ccRCC molecular subgroup 3 -> randomisation: TKI (sunitinib 50mg daily or Pazopanib 800mg daily) according to investigator's choice until disease progression, unacceptable toxicity or other reasons specified in the protocol.
  Interventions: Drug: Pazopanib; Drug: Sunitinib

INTERVENTIONS:
Drug: Nivolumab — For Arms 1A and 4A:
  Nivolumab alone administered IV over 60 minutes at 240 mg every 2 weeks until disease progression, unacceptable toxicity or other reasons specified in the protocol.
  For Arms 1B, 2B, 3B and 4B:
  Nivolumab administered IV over 60 minutes at 3 mg/kg combined with ipilimumab administered IV over 30 minutes at 1 mg/kg every 3 weeks for 4 doses followed by nivolumab administered IV over 60 minutes at 240 mg every 2 weeks until disease progression, unacceptable toxicity or other reasons specified in the protocol.
  Starting from the Cycle 7 possibility to switch from nivolumab 240 mg every 2 weeks to 480 mg every 4 weeks according to the Investigator's preference.
  Other Names: BMS-936558; Opdivo
  Arms: ccRCC molecular subgroup 1: 1A; ccRCC molecular subgroup 1: 1B; ccRCC molecular subgroup 2: 2B; ccRCC molecular subgroup 3: 3B; ccRCC molecular subgroup 4: 4A; ccRCC molecular subgroup 4: 4B
Drug: Ipilimumab — For Arms 1B, 2B, 3B and 4B:
  Ipilimumab administered IV over 30 minutes at 1 mg/kg every 3 weeks combined with Nivolumab administered IV over 60 minutes at 3 mg/kg for 4 doses until disease progression, unacceptable toxicity or other reasons specified in the protocol.
  Other Names: YERVOY; BMS-734016
  Arms: ccRCC molecular subgroup 1: 1B; ccRCC molecular subgroup 2: 2B; ccRCC molecular subgroup 3: 3B; ccRCC molecular subgroup 4: 4B
Drug: Pazopanib — For Arms 2C and 3C (TKI pazopanib or sunitinib):
  Pazopanib 800 mg orally QD until disease progression, unacceptable toxicity or other reasons specified in the protocol
  Other Names: Votrient
  Arms: ccRCC molecular subgroup 2: 2C; ccRCC molecular subgroup 3: 3C
Drug: Sunitinib — For Arms 2C and 3C (TKI pazopanib or sunitinib):
  Sunitinib 50 mg orally QD until disease progression, unacceptable toxicity or other reasons specified in the protocol
  Other Names: Sutent
  Arms: ccRCC molecular subgroup 2: 2C; ccRCC molecular subgroup 3: 3C

SUMMARY:
Disease and Stage: naïve metastatic kidney cancer.

A multicenter, randomized, a Phase 2 BIOmarker driven trial with Nivolumab and Ipilimumab or VEGFR tKi in naïve metastatic Kidney cancer

DETAILED DESCRIPTION:
Research Hypothesis: Molecular groups of ccrcc will define patients who will respond to nivolumab alone, nivolumab combined with ipilimumab, or VEGFR-TKI (sunitinib or pazopanib) in subjects with previously untreated metastatic renal cell carcinoma (mRCC).

Conditions:

* Advanced or metastatic RCC: previously untreated in metastatic setting.
* Frozen tumor samples available for molecular group determination.
* Determination of molecular subgroup prior to randomization.

Product(s):

* ARM A: nivolumab alone administered IV over 60 minutes at 240 mg every 2 weeks (molecular group 1 and 4).
* ARM B : Nivolumab administered IV over 60 minutes at 3 mg/kg combined with ipilimumab administered IV over 30 minutes at 1 mg/kg every 3 weeks for 4 doses followed by nivolumab administered IV over 60 minutes at 240 mg every 2 weeks

starting from the Cycle 7 possibility to switch from nivolumab 240 mg every 2 weeks to 480 mg every 4 weeks according to the Investigator's preference (Arm A and B),

- ARM C: TKI (molecular group 2 and 3), pazopanib or sunitinib according to investigator's choice until disease progression, unacceptable toxicity or other reasons specified in the protocol.

Biological assessments:

Molecular groups (1 to 4) will be determined for all patients from frozen tumor tissue samples or from fresh tumor samples immediately stored in "RNA later" medium.

Further exploratory biological assessments will be performed in order to define predictive biomarkers of response to N+I, N alone or TKI (sunitinib or pazopanib) by analyzing tumor specimens and blood samples:

* To assess gene expression of immune population markers in the primary tumor as well as in the metastases before beginning treatment, and at progression if safely achievable.
* Gene expression analysis will be performed from frozen and FFPE tumor tissue in order to compare the two methods.
* To assess the density and phenotype of selected immune populations (CD8, CD3/CD20, PD-1, TIM-3, LAG3, FoxP3) as well as the phenotype of tumor cells (PD-L1, PD-L2) by immunohistochemistry (IHC) in the primary tumor and metastases, before treatment initiation and at progression if safely achievable.
* To assess the functional status of peripheral blood lymphocytes (PBL) by flow cytometry, before treatment initiation, during treatment, and at progression.
* To quantify plasmatic angiogenesis-related (i.e. VEGF-A, VEGF-C its soluble receptors VEGFR-1 and 2 and co-receptors neuropilin 1 and 2, angiopoietins, SDF-1, PDGFs…)) and endothelial cell-derived molecules (i.e. endoglin, VE-cadherin) before treatment initiation, during treatment, and at progression.
* To correlate plasmatic angiogenesis-related molecules with tumor vascularization studied by immunofluorescence (IF) and a multi-spectral analyzer (Vectra technology) on tumor tissue.
* To investigate a predictive role of the response of CXCL7 and sCD146 to TKI, nivolumab and/or nivolumab+ipilimumab.
* To determine whether the mutation and methylation analysis of circulating tumor DNA can be used as predictive biomarker of response, resistance to treatment or progression.
* Identify genetic and epigenetic alterations associated with either response or resistance to immune checkpoint inhibitors and tyrosine kinase inhibitors
* Evaluate association between immune cells composing tumor microenvironment and response and/or resistance to immune checkpoint inhibitors or tyrosine kinase inhibitors
* Evaluate additional genetic and epigenetic tumor alterations at resistance/progression or after resection of residual mass.

Statistical Considerations:

An adaptative design will be used to ensure that conclusions can be made with a limited number of patients in each molecular group, which is the major constraint of the study.

Sample Size: Approximately 150 patients are planned to be treated. Given an expected failure rate of molecular grouping of less than 20%, 150-200 patients must be included.

ELIGIBILITY:
Key Inclusion Criteria:

* Histological confirmation of RCC with a clear-cell component. Patients with TFE3 or TFEB translocation proven by cytogenetic analysis or by fluorescence in situ hybridization (FISH) are eligible.
* Metastatic (American Joint Committee on Cancer [AJCC] Stage IV) RCC
* No prior systemic therapy for mRCC
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤2
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Frozen tumor samples (primary tumor and/or metastasis biopsies) must be available and received by the central laboratory (Cordelier Research Center) to determine molecular groups. (Note: fine needle aspiration [FNA] and bone metastases samples are not acceptable for submission).
* Molecular group has to be determined prior to randomization.
* Formalin-fixed, paraffin-embedded (FFPE) tumor tissue available for biomarker (gene expression and immunohistochemistry (IHC)) analysis.

Key Exclusion Criteria:

* Any untreated CNS metastases. Patients with CNS metastases will be eligible if they are: asymptomatic, without significant oedema, not on corticosteroids, not eligible for radiation therapy/surgery or have already received radiation therapy.
* Prior systemic treatment with vascular endothelial growth factor (VEGF) or VEGF receptor-targeted therapy (including, but not limited to, sunitinib, pazopanib, axitinib, tivozanib, and bevacizumab) except in an adjuvant setting with a free interval of more than 1 year.
* Prior treatment with an anti-programmed cell death protein 1 (PD-1), anti-programmed death-ligand 1 (PD-L1), anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids (>10 mg daily prednisone equivalent) or immunosuppressive medications except for syndromes which would not be expected to recur in the absence of an external trigger. Subjects with vitiligo or type 1 diabetes mellitus or residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement are permitted to enroll.
* Any condition requiring systemic treatment with corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroid doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Uncontrolled adrenal insufficiency.
* Ongoing symptomatic cardiac dysrhythmias, uncontrolled atrial fibrillation, or prolongation of the Fridericia corrected QT (QTcF) interval defined as >450 msec for males and >470 msec for females, where QTcF = QT / 3√RR.
* Poorly controlled hypertension (defined as systolic blood pressure (SBP) of >150 mmHg or diastolic blood pressure (DBP) of >90 mmHg), despite antihypertensive therapy.
* History of any of the following cardiovascular conditions within 12 months of enrollment: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery by-pass graft surgery, symptomatic peripheral vascular disease, class III or IV congestive heart failure, as defined by the New York Heart Association.
* History of cerebrovascular accident including transient ischemic attack within the past 12 months.
* History of deep vein thrombosis (DVT) unless adequately treated with low molecular weight heparin.
* History of pulmonary embolism within the past 6 months unless stable, asymptomatic, and treated with low molecular weight heparin for at least 6 weeks.
* Known history of COPD (of any stage).
* Known history of uveitis or complaint of double vision.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months.
* Serious, non-healing wound or ulcer.
* Evidence of active bleeding or bleeding susceptibility; or medically significant hemorrhage within prior 30 days.
* Any requirement for anti-coagulation, except for low molecular weight heparin.
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Any positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection.
* Known medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the Investigator's opinion, would increase the risk associated with study participation or study drug administration, or interfere with the interpretation of safety results.
* Known history of hyperesthesia, hypoesthesia, paresthesia, dysesthesia, peripheral motor neuropathy, peripheral sensory, neuropathy, and polyneuropathy.
* Major surgery (e.g., nephrectomy) less than 35 days prior to the first dose of study drug.
* Focal radiation therapy less than 14 days prior to the first dose of study drug.
* Receiving concomitant CYP3A4 inducers or strong CYP3A4 inhibitors
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of cabozantinib (e.g., malabsorptive disorder, ulcerative disease, uncontrolled nausea, vomiting, diarrhea, or small bowel resection).
* Any of the following laboratory test findings:

  1. WBC <2,000/mm3
  2. Hemoglobin ≤9.0 g/dL
  3. Neutrophils <1,500/mm3
  4. Platelets <100,000/mm3
  5. AST or ALT >3 x ULN (>5 x ULN if liver metastases are present)
  6. Lipase and amylase > 1.5 ULN
  7. Total Bilirubin >1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin <3.0 mg/dL)
  8. Serum creatinine >1.5 x ULN or creatinine clearance <40 mL/min (measured or calculated by Cockroft-Gault formula)
  9. Proteinuria: patients with ≥2+ protein on urine dipstick at baseline must undergo a 24-hour urine collection for protein then if > 1.0 g of protein patient will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
ORR evaluation according to molecular groups (ccRCC1 to 4) and assigned treatment | 54 months
  ORR evaluation according to molecular groups (ccRCC1 to 4) and assigned treatment (nivolumab monotherapy, nivolumab combined with ipilimumab, or TKI: sunitinib or pazopanib), based on Investigator assessments.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 54 months
  progression-free survival (PFS) in subjects with previously untreated mRCC according to molecular groups and assigned treatment, based on Investigator radiological assessments.
Overall Survival | 54 months
  To evaluate OS in subjects with previously untreated mRCC according to molecular groups and assigned treatment.
Objective response rate at 22 weeks | at 22 weeks
  To evaluate objective response rate at 22 weeks as a surrogate of other endpoints according to molecular groups and assigned treatment.
Duration of treatment (DOT) | 54 months
  To evaluate the duration of treatment (DOT) of nivolumab combined with ipilimumab or nivolumab alone or cabozantinib in subjects with previously untreated mRCC according to their molecular subgroup (1&4 vs 2&3).
Duration of response (DOR) | 54 months
  To evaluate the duration of response (DOR) of nivolumab combined with ipilimumab or nivolumab alone or cabozantinib in subjects with previously untreated mRCC according to their molecular subgroup (1&4 vs 2&3).
Number of Participants With Treatment-Related Adverse Events | 54 months
  To estimate the incidence of AEs associated with nivolumab combined with ipilimumab or nivolumab alone or cabozantinib in all treated subjects with previously untreated mRCC.
Gene expression of immune population markers | at baseline at progression (36 months maximum)
  To assess gene expression of immune population markers in the primary tumor as well as in the metastases before beginning treatment, and at progression if safely achievable.populations (CD3, CD8...) and regulatory markers (PD-1, LAG-3…) within the primary tumor, and metastases whenever possible, using frozen and FFPE tumor tissue.
Gene expression levels obtained from FFPE | at the end of the study (36 months)
  Gene expression levels obtained from FFPE tumor tissue (exploratory method) will be compared to those obtained with frozen tumor tissue (standard method).
Functional status of peripheral blood lymphocytes (PBL) | at baseline, at cycle 2 and at progression (36 months maximum)
  To assess the functional status of peripheral blood lymphocytes (PBL) by flow cytometry, before treatment initiation, during treatment, and at progression.
Association between non-immune tissue and circulating biomarkers and outcomes | 36 months maximum
  To explore the association between non-immune tissue and circulating biomarkers and outcomes (ORR, ORR at 22 weeks, OS and PFS).
Mutation and methylation analysis of circulating tumor DNA | 36 months maximum
  The initial rate of ctDNA and its evolution will be correlated to the clinical evolution of patients and progression-free survival.
Genetic and epigenetic alterations | 36 months maximum
  To identify genetic and epigenetic alterations associated with either response or resistance to immune checkpoint inhibitors and tyrosine kinase inhibitors.
association between immune cells composing tumor microenvironment and response and/or resistance | 36 months maximum
  To evaluate the association between immune cells composing tumor microenvironment and response and/or resistance to immune checkpoint inhibitors or tyrosine kinase inhibitors.
additional genetic and epigenetic tumor alterations | 36 months maximum
  To evaluate additional genetic and epigenetic tumor alterations at resistance/progression or after resection of residual mass.

CONTACTS AND LOCATIONS:
Overall Officials: Yann-Alexandre VANO, MD, Principal Investigator — Hôpital Européen Georges Pompidou; Oncology department of Pr Stéphane OUDARD
Locations (16):
- France (16):
  - Hôpital Saint André, CHU de Bordeaux, Bordeaux
  - Centre Francois Baclesse, Caen
  - CHU Henri-Mondor, Créteil
  - Centre OSCAR LAMBRET LILLE, Lille
  - Institut Paoli Calmettes (IPC), Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut de Cancérologie du Gard - CHU Caremeau, Nîmes
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Cochin, Paris
  - Centre Hospitalier Lyon Sud - Institut de Cancérologie des Hospices Civils de Lyon (IC-HCL), Pierre-Bénite
  - Centre Eugene Marquis, Rennes
  - Hôpitaux universitaires de Strasbourg, Strasbourg
  - Hopital Foch, Suresnes
  - Institut Claudius Regaud, Toulouse
  - CHU Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davidson G, Helleux A, Vano YA, Lindner V, Fattori A, Cerciat M, Elaidi RT, Verkarre V, Sun CM, Chevreau C, Bennamoun M, Lang H, Tricard T, Fridman WH, Sautes-Fridman C, Su X, Plassard D, Keime C, Thibault-Carpentier C, Barthelemy P, Oudard SM, Davidson I, Malouf GG. Mesenchymal-like Tumor Cells and Myofibroblastic Cancer-Associated Fibroblasts Are Associated with Progression and Immunotherapy Response of Clear Cell Renal Cell Carcinoma. Cancer Res. 2023 Sep 1;83(17):2952-2969. doi: 10.1158/0008-5472.CAN-22-3034. PMID 37335139
- [Derived] Vano YA, Elaidi R, Bennamoun M, Chevreau C, Borchiellini D, Pannier D, Maillet D, Gross-Goupil M, Tournigand C, Laguerre B, Barthelemy P, Coquan E, Gravis G, Houede N, Cancel M, Huillard O, Beuzeboc P, Fournier L, Mejean A, Cathelineau X, Doumerc N, Paparel P, Bernhard JC, de la Taille A, Bensalah K, Tricard T, Waeckel T, Pignot G, Braychenko E, Caruso S, Sun CM, Verkarre V, Lacroix G, Moreira M, Meylan M, Bougouin A, Phan L, Thibault-Carpentier C, Zucman-Rossi J, Fridman WH, Sautes-Fridman C, Oudard S. Nivolumab, nivolumab-ipilimumab, and VEGFR-tyrosine kinase inhibitors as first-line treatment for metastatic clear-cell renal cell carcinoma (BIONIKK): a biomarker-driven, open-label, non-comparative, randomised, phase 2 trial. Lancet Oncol. 2022 May;23(5):612-624. doi: 10.1016/S1470-2045(22)00128-0. Epub 2022 Apr 4. PMID 35390339
- [Derived] Epaillard N, Simonaggio A, Elaidi R, Azzouz F, Braychenko E, Thibault C, Sun CM, Moreira M, Oudard S, Vano YA. BIONIKK: A phase 2 biomarker driven trial with nivolumab and ipilimumab or VEGFR tyrosine kinase inhibitor (TKI) in naive metastatic kidney cancer. Bull Cancer. 2020 Jun;107(5S):eS22-eS27. doi: 10.1016/S0007-4551(20)30283-6. PMID 32620212